CLINICAL TRIAL: NCT04062708
Title: CHIO3 Trial: CHemotherapy Combined With Immune Checkpoint Inhibitor for Operable Stage IIIA/B Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-46
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
Keywords: Stage IIIA/IIIB (T1-3,N2) Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Combined neoadjuvant platinum doublet chemotherapy plus durvalumab followed by surgery, postoperative radiation and adjuvant durvalumab for 13 cycles.
  Interventions: Drug: Durvalumab; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab — Preoperative Treatment:
  * Non-squamous NSCLC: durvalumab 1125 mg, followed by pemetrexed 500 mg/m2 IV with cisplatin 75 mg/m2 IV, every 3 weeks, for 4 cycles
  * Squamous NSCLC: durvalumab 1125 mg, followed by docetaxel 75 mg/m2 IV with cisplatin 75 mg/m2 IV, every 3 weeks, for 4 cycles
  Adjuvant Therapy:
  • 1-6 weeks after completion of radiotherapy, durvalumab 1500 mg IV every 4 weeks will be administered for 13 cycles.
  Other Names: Imfinzi
Procedure: Surgery — Patients will be re-evaluated following preoperative treatment to assess if patient is still medically fit to withstand surgery. Eligible patients will then undergo lobectomy, bilobectomy, sleeve lobectomy or other extended resection, or a pneumonectomy will be performed at the discretion of the attending thoracic surgeon.
Radiation: Radiotherapy — 4-10 weeks after surgery, patients will receive 54 Gy of radiotherapy with single daily fractions.

SUMMARY:
This is a single arm, phase II trial of combined neoadjuvant platinum doublet chemotherapy plus durvalumab followed by surgery, postoperative radiation and adjuvant durvalumab for 13 cycles for patients with potentially resectable stage IIIA and IIIB (T1-3, N2) NSCLC (per the 8th International Association for the Study of Lung Cancer classification). The primary objective of this study is to increase N2 nodal clearance (N2NC) to 50% or greater for combined platinum doublet chemotherapy with durvalumab induction therapy from historical rate of 30% for platinum doublet chemotherapy alone in patients with potentially resectable stage IIIA/B (N2) NSCLC.

DETAILED DESCRIPTION:
In the preoperative period, patients who have undergone adequate mediastinal evaluation and are considered operable will be treated with durvalumab 1125 mg IV every 3 weeks (Q3W) in combination with platinum doublet chemotherapy (cisplatin with pemetrexed or docetaxel, depending upon histology).

Patients will undergo postoperative radiation (54Gy) within 4-10 weeks after surgery (unless single station N2 at registration with resultant ypT0N0 after neoadjuvant therapy).

One to 6 weeks after completion of radiation, patients will receive adjuvant durvalumab 1500 mg IV every 4weeks (Q4W) for 1 year.

Patients who do not have surgery due to refusal, physician decision, or local and distant progression will have to discontinue study treatment.

All participants will have imaging assessment prior to surgery after Cycle 2 (Week 6) and after Cycle 4 (Weeks 13 15). Patients will undergo potentially curable surgery as per standard of care.

Patients will undergo imaging assessment every 12 weeks after surgery for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Operability Criteria:

1. ECOG Performance Status 0-1.
2. Absence of major associated comorbidities that increase the surgery risk to an unacceptable level.
3. Pulmonary function capacity capable of tolerating the proposed lung resection. FEV1 at least 2 L. If less than 2 L, the predicted postoperative forced expiratory volume in 1 second (FEV1) must be >0.8 L or be >35% of the predicted value. Postoperative predicted DLCO ≥35% is required.

Inclusion Criteria:

1. Patients who are at least 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
3. Life expectancy of at least 12 weeks.
4. Patients with potentially resectable IIIA/B (T1-3, N2) NSCLC (per the 8th International Association for the Study of Lung Cancer classification) who are candidates for surgery with intent of R0 resection. Invasive T3 disease (eg, phrenic nerve, pericardium, chest wall other than Pancoast superior sulcus) may be included if the surgeon and study team deem it to be resectable. T4 disease per AJCC 8th edition staging system is excluded given the lack of benefit of surgery in T4N2.
5. Patients must be evaluated by a thoracic surgeon within 4 weeks of registration.
6. Operability is defined as having adequate pulmonary, cardiac, renal, nutritional, musculoskeletal, neurologic, and cognitive capacity to undergo major pulmonary resection with acceptable morbidity and mortality.
7. N2 nodes must be discrete (ie, not invading surrounding structures) and less than 3 cm in maximum diameter.
8. Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
9. Pathologically proven N2 disease within 4 weeks of registration. PET/CT positivity in the ipsilateral mediastinal nodes will not be sufficient to establish N2 nodal status. Mediastinal lymph node sampling biopsy is required pre-operatively by at least one of the following:

   * Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA);
   * Mediastinoscopy;
   * Mediastinotomy (Chamberlain procedure);
   * Endoscopic ultrasound guided node aspiration (EUS);
   * Video-assisted thoracoscopy; OR
   * Fine needle aspiration by image guidance.
   * Endobronchial ultrasound (EBUS) or mediastinoscopy or other tissue sampling (at least 2 stations must be biopsied, with at least one station positive for N2 disease). If there are any mediastinal nodes suspicious by CT (>1.5 cm) or PET in N3 stations, they must be biopsied. If biopsy proven involvement in an N3 station, the patient is excluded.
10. Mediastinal nodal biopsy or aspiration can only be omitted in the special circumstance in which ALL of the following are true:

    * The tumor is left sided;
    * The only mediastinal nodal involvement is a node visible in the AP (level 5) region on CT scan;
    * Distinct primary tumor separate from the nodes; AND
    * Biopsy proven non-small cell histology from the primary tumor.
11. No prior history of thoracic radiation.
12. Organ and marrow function definitions (example below)

    * leukocytes ≥3,000/mcL
    * absolute neutrophil count ≥1,500/mcL
    * platelets ≥100,000/mcL
    * Hemoglobin >9.0 g/dL
    * total bilirubin within normal institutional limits
    * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
    * creatinine within normal institutional limits OR
    * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
13. Patients are capable of giving informed consent and/or have an acceptable surrogate capable of giving consent on the subject's behalf.
14. Nonpregnant and non-nursing. The effect of durvalumab on the fetus is unknown.
15. Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 3 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses >1 year.
16. Evidence of postmenopausal status or negative urinary or serum pregnancy test for female premenopausal patients. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
17. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
18. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 12 weeks after the last dose of study therapy.

Exclusion Criteria:

1. Any prior treatment for NSCLC.
2. Prior thoracic radiation.
3. Patients with ≥Grade 2 peripheral neuropathy.
4. Any active or history of autoimmune disease (including any history of inflammatory bowel disease) or history of a syndrome that required systemic steroids or immunosuppressive medications, except for patients with vitiligo or resolved childhood asthma/atopy.
5. Patients requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Patients with previous malignancies (except nonmelanoma skin cancers, in situ bladder, gastric, breast, colon or cervical cancers/dysplasia) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
7. History of solid organ transplant.
8. N3 nodal disease.
9. Mixed small cell/NSCLC will be excluded.
10. Pregnant or breastfeeding.
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], active diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia.
    * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
    * Any chronic skin condition that does not require systemic therapy.
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
    * Patients with celiac disease controlled by diet alone.
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
N2 nodal clearance (N2NC) | 5 years
  To increase N2 nodal clearance (N2NC) to 50% or greater for combined platinum doublet chemotherapy with durvalumab induction from an historical rate of 30% for platinum doublet chemotherapy alone in patients with potentially resectable stage IIIA/B (N2) NSCLC.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  To evaluate the safety and tolerability of neoadjuvant platinum doublet chemotherapy and durvalumab followed by surgery followed by adjuvant radiation and durvalumab.
Radiographic response rate | 5 years
  To assess the radiographic response rate of neoadjuvant platinum doublet chemotherapy and durvalumab.
Rate of major pathologic response and pathologic complete response | 16 weeks
  To evaluate the rate of major pathologic response and pathologic complete response in the resected primary tumor and lymph nodes following neoadjuvant combination therapy.
Evaluate event free survival (EFS) | 5 years
  EFS evaluated from the time of registration to one of the following events, whichever comes first: a) radiographic disease progression, b) local progression as defined by lymph node progression precluding surgery, c) inability to resect the tumor, d) local or distant recurrence, e) death due to any cause.
Overall survival rate | 5 years
  To evaluate overall survival rate from the time of registration
Rate of complete resection. | 16 weeks
  To assess the rate of complete resection.
Post-operative complications | Within 30 days of surgery
  To assess post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Linda Martin, MD, MPH, Study Chair — University of Virginia; Jyoti Patel, MD, Study Chair — University of Chicago; James Urbanic, MD, Study Chair — University of California, San Diego; David Kozono, MD, Study Director — Alliance Foundation Trials, LLC.
Locations (9):
- United States (9):
  - NorthWestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York
  - Baptist Cancer Center, Memphis, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Darling GE, Li F, Patsios D, Massey C, Wallis AG, Coate L, Keshavjee S, Pierre A, De Perrot M, Yasufuku K, Cypel M, Waddell T. Neoadjuvant chemoradiation and surgery improves survival outcomes compared with definitive chemoradiation in the treatment of stage IIIA N2 non-small-cell lung cancer. Eur J Cardiothorac Surg. 2015 Nov;48(5):684-90; discussion 690. doi: 10.1093/ejcts/ezu504. Epub 2015 Jan 6. PMID 25567960
- [Background] Pless M, Stupp R, Ris HB, Stahel RA, Weder W, Thierstein S, Gerard MA, Xyrafas A, Fruh M, Cathomas R, Zippelius A, Roth A, Bijelovic M, Ochsenbein A, Meier UR, Mamot C, Rauch D, Gautschi O, Betticher DC, Mirimanoff RO, Peters S; SAKK Lung Cancer Project Group. Induction chemoradiation in stage IIIA/N2 non-small-cell lung cancer: a phase 3 randomised trial. Lancet. 2015 Sep 12;386(9998):1049-56. doi: 10.1016/S0140-6736(15)60294-X. Epub 2015 Aug 11. PMID 26275735
- [Background] Higgins K, Chino JP, Marks LB, Ready N, D'Amico TA, Clough RW, Kelsey CR. Preoperative chemotherapy versus preoperative chemoradiotherapy for stage III (N2) non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1462-7. doi: 10.1016/j.ijrobp.2009.01.069. Epub 2009 May 19. PMID 19467798
- [Background] Edelman MJ, Hu C, Le QT, Donington JS, D'Souza WD, Dicker AP, Loo BW, Gore EM, Videtic GMM, Evans NR, Leach JW, Diehn M, Feigenberg SJ, Chen Y, Paulus R, Bradley JD. Randomized Phase II Study of Preoperative Chemoradiotherapy +/- Panitumumab Followed by Consolidation Chemotherapy in Potentially Operable Locally Advanced (Stage IIIa, N2+) Non-Small Cell Lung Cancer: NRG Oncology RTOG 0839. J Thorac Oncol. 2017 Sep;12(9):1413-1420. doi: 10.1016/j.jtho.2017.06.007. Epub 2017 Jun 16. PMID 28629896
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Postoperative radiotherapy in non-small-cell lung cancer: systematic review and meta-analysis of individual patient data from nine randomised controlled trials. PORT Meta-analysis Trialists Group. Lancet. 1998 Jul 25;352(9124):257-63. PMID 9690404
- [Background] Dautzenberg B, Arriagada R, Chammard AB, Jarema A, Mezzetti M, Mattson K, Lagrange JL, Le Pechoux C, Lebeau B, Chastang C. A controlled study of postoperative radiotherapy for patients with completely resected nonsmall cell lung carcinoma. Groupe d'Etude et de Traitement des Cancers Bronchiques. Cancer. 1999 Jul 15;86(2):265-73. doi: 10.1002/(sici)1097-0142(19990715)86:23.0.co;2-b. PMID 10421262
- [Background] Debevec M, Bitenc M, Vidmar S, Rott T, Orel J, Strojan P, Kovac V. Postoperative radiotherapy for radically resected N2 non-small-cell lung cancer (NSCLC): randomised clinical study 1988-1992. Lung Cancer. 1996 Feb;14(1):99-107. doi: 10.1016/0169-5002(95)00515-3. PMID 8696724
- [Background] Stephens RJ, Girling DJ, Bleehen NM, Moghissi K, Yosef HM, Machin D. The role of post-operative radiotherapy in non-small-cell lung cancer: a multicentre randomised trial in patients with pathologically staged T1-2, N1-2, M0 disease. Medical Research Council Lung Cancer Working Party. Br J Cancer. 1996 Aug;74(4):632-9. doi: 10.1038/bjc.1996.413. PMID 8761382
- [Background] Burdett S, Rydzewska L, Tierney J, Fisher D, Parmar MK, Arriagada R, Pignon JP, Le Pechoux C; PORT Meta-analysis Trialists Group. Postoperative radiotherapy for non-small cell lung cancer. Cochrane Database Syst Rev. 2016 Oct 11;10(10):CD002142. doi: 10.1002/14651858.CD002142.pub4. PMID 27727451
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Suntharalingam M, Paulus R, Edelman MJ, Krasna M, Burrows W, Gore E, Wilson LD, Choy H. Radiation therapy oncology group protocol 02-29: a phase II trial of neoadjuvant therapy with concurrent chemotherapy and full-dose radiation therapy followed by surgical resection and consolidative therapy for locally advanced non-small cell carcinoma of the lung. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):456-63. doi: 10.1016/j.ijrobp.2011.11.069. Epub 2012 Apr 28. PMID 22543206
- [Background] Jaklitsch MT, Herndon JE 2nd, DeCamp MM Jr, Richards WG, Kumar P, Krasna MJ, Green MR, Sugarbaker DJ. Nodal downstaging predicts survival following induction chemotherapy for stage IIIA (N2) non-small cell lung cancer in CALGB protocol #8935. J Surg Oncol. 2006 Dec 1;94(7):599-606. doi: 10.1002/jso.20644. PMID 17039491
- [Background] Betticher DC, Hsu Schmitz SF, Totsch M, Hansen E, Joss C, von Briel C, Schmid RA, Pless M, Habicht J, Roth AD, Spiliopoulos A, Stahel R, Weder W, Stupp R, Egli F, Furrer M, Honegger H, Wernli M, Cerny T, Ris HB. Mediastinal lymph node clearance after docetaxel-cisplatin neoadjuvant chemotherapy is prognostic of survival in patients with stage IIIA pN2 non-small-cell lung cancer: a multicenter phase II trial. J Clin Oncol. 2003 May 1;21(9):1752-9. doi: 10.1200/JCO.2003.11.040. PMID 12721251
- [Background] Thomas M, Rube C, Hoffknecht P, Macha HN, Freitag L, Linder A, Willich N, Hamm M, Sybrecht GW, Ukena D, Deppermann KM, Droge C, Riesenbeck D, Heinecke A, Sauerland C, Junker K, Berdel WE, Semik M; German Lung Cancer Cooperative Group. Effect of preoperative chemoradiation in addition to preoperative chemotherapy: a randomised trial in stage III non-small-cell lung cancer. Lancet Oncol. 2008 Jul;9(7):636-48. doi: 10.1016/S1470-2045(08)70156-6. Epub 2008 Jun 24. PMID 18583190
- [Background] Ripley RT, Suzuki K, Tan KS, Adusumilli PS, Huang J, Park BJ, Downey RJ, Rizk NP, Rusch VW, Bains M, Jones DR. Postinduction positron emission tomography assessment of N2 nodes is not associated with ypN2 disease or overall survival in stage IIIA non-small cell lung cancer. J Thorac Cardiovasc Surg. 2016 Apr;151(4):969-77, 979.e1-3. doi: 10.1016/j.jtcvs.2015.09.127. Epub 2015 Oct 19. PMID 26614420
- [Background] van Meerbeeck JP, Kramer GW, Van Schil PE, Legrand C, Smit EF, Schramel F, Tjan-Heijnen VC, Biesma B, Debruyne C, van Zandwijk N, Splinter TA, Giaccone G; European Organisation for Research and Treatment of Cancer-Lung Cancer Group. Randomized controlled trial of resection versus radiotherapy after induction chemotherapy in stage IIIA-N2 non-small-cell lung cancer. J Natl Cancer Inst. 2007 Mar 21;99(6):442-50. doi: 10.1093/jnci/djk093. PMID 17374834
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] De Leyn P, Dooms C, Kuzdzal J, Lardinois D, Passlick B, Rami-Porta R, Turna A, Van Schil P, Venuta F, Waller D, Weder W, Zielinski M. Revised ESTS guidelines for preoperative mediastinal lymph node staging for non-small-cell lung cancer. Eur J Cardiothorac Surg. 2014 May;45(5):787-98. doi: 10.1093/ejcts/ezu028. Epub 2014 Feb 26. PMID 24578407
- [Background] Chapet O, Kong FM, Quint LE, Chang AC, Ten Haken RK, Eisbruch A, Hayman JA. CT-based definition of thoracic lymph node stations: an atlas from the University of Michigan. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):170-8. doi: 10.1016/j.ijrobp.2004.12.060. PMID 16111586
- [Background] Kong FM, Ritter T, Quint DJ, Senan S, Gaspar LE, Komaki RU, Hurkmans CW, Timmerman R, Bezjak A, Bradley JD, Movsas B, Marsh L, Okunieff P, Choy H, Curran WJ Jr. Consideration of dose limits for organs at risk of thoracic radiotherapy: atlas for lung, proximal bronchial tree, esophagus, spinal cord, ribs, and brachial plexus. Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1442-57. doi: 10.1016/j.ijrobp.2010.07.1977. Epub 2010 Oct 8. PMID 20934273
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009 Sep;49(9):1012-24. doi: 10.1177/0091270009337512. Epub 2009 Jul 20. PMID 19620385
- [Background] Zhang S, Shi R, Li C, Parivar K, Wang DD. Fixed dosing versus body size-based dosing of therapeutic peptides and proteins in adults. J Clin Pharmacol. 2012 Jan;52(1):18-28. doi: 10.1177/0091270010388648. Epub 2011 Jan 13. PMID 21233304
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Brahmer JR, Lacchetti C, Thompson JA. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline Summary. J Oncol Pract. 2018 Apr;14(4):247-249. doi: 10.1200/JOP.18.00005. Epub 2018 Mar 8. No abstract available. PMID 29517954
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Rustin GJ, Quinn M, Thigpen T, du Bois A, Pujade-Lauraine E, Jakobsen A, Eisenhauer E, Sagae S, Greven K, Vergote I, Cervantes A, Vermorken J. Re: New guidelines to evaluate the response to treatment in solid tumors (ovarian cancer). J Natl Cancer Inst. 2004 Mar 17;96(6):487-8. doi: 10.1093/jnci/djh081. No abstract available. PMID 15026475
- [Background] Bubley GJ, Carducci M, Dahut W, Dawson N, Daliani D, Eisenberger M, Figg WD, Freidlin B, Halabi S, Hudes G, Hussain M, Kaplan R, Myers C, Oh W, Petrylak DP, Reed E, Roth B, Sartor O, Scher H, Simons J, Sinibaldi V, Small EJ, Smith MR, Trump DL, Wilding G, et al. Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol. 1999 Nov;17(11):3461-7. doi: 10.1200/JCO.1999.17.11.3461. PMID 10550143
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Vergote I, Rustin GJ, Eisenhauer EA, Kristensen GB, Pujade-Lauraine E, Parmar MK, Friedlander M, Jakobsen A, Vermorken JB. Re: new guidelines to evaluate the response to treatment in solid tumors [ovarian cancer]. Gynecologic Cancer Intergroup. J Natl Cancer Inst. 2000 Sep 20;92(18):1534-5. doi: 10.1093/jnci/92.18.1534. No abstract available. PMID 10995813